CLINICAL TRIAL: NCT02972879
Title: Effectiveness of Non-surgical Interventions for the Trigger Finger: a Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beatriz Sernajoto Cristiani Pedro (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Sponsor-Investigator, Beatriz Sernajoto Cristiani Pedro, BSCPedro, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSCPedro
Record Dates: First submitted 2016-11-07; First posted 2016-11-25 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Trigger Finger
Keywords: trigger finger; Therapeutic Modalities; Corticosteroid Injection; non-surgical treatment; physical therapy
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Modalities (Active Comparator): * Group 1: Metal orthotic, keeping 0º of the extension of the proximal interphalangeal joint, during all day, for 5 weeks, stopping the use only for bathing
  * Group 2: 10 LLLT sessions applications on the A1 pulley and lump formed on the flexor tendon of the the affected finger; Two sessions per week, five weeks of treatment.
  * Group 3: Paraffin bath 2 times a week for 20 minutes (total of 10 sessions).
  Interventions: Procedure: Therapeutic modalities: Orthotic (Group 1); Procedure: Therapeutic modalities: LLLT (Group 2); Procedure: Therapeutic modalities: Paraffin (Group 3)
- Corticosteroid injection (Active Comparator): Group 4: Corticosteroid injection in the A1 pulley, 1 application.
  Interventions: Procedure: Corticosteroid injection (Group 4)

INTERVENTIONS:
Procedure: Therapeutic modalities: Orthotic (Group 1) — participants will be instructed to remove the orthosis only two hours in the morning, two hours in the afternoon and two hours at night to avoid joint stiffness
  Other Names: Metal orthotic
  Arms: Therapeutic Modalities
Procedure: Therapeutic modalities: LLLT (Group 2) — The LLLT parameters are:
  * LASER 904nm
  * P: 1.5W/cm²
  * 30mV/cm²
  * Area 2 cm²
  * 1 Joule por ponto ( in the A1 pulley)
  Other Names: Ibramed's LASERPULSED 904nm
  Arms: Therapeutic Modalities
Procedure: Therapeutic modalities: Paraffin (Group 3) — Paraffin will be heated and maintained at 50 ° C. Participants will immerse their affected hand 10 times in heated paraffin, then they will roll up their affected hand in a towel that they will bring, after 20 minutes timed by a trained professional, the subjects will remove the towel and "paraffin glove":
  Other Names: Bath Paraffin Carci´s
  Arms: Therapeutic Modalities
Procedure: Corticosteroid injection (Group 4) — The injection solution is composed of 1 ml of betamethasone and 1 ml of 2% lidocaine.This group may repeat the procedure in two weeks if they report that there was no improvement of the triggering or pain.
  Other Names: Bethametasone
  Arms: Corticosteroid injection

SUMMARY:
The aim of this study is to assess the effectiveness of therapeutic modalities (paraffin, ultrasound and orthotics) versus corticosteroid injection for trigger finger.

DETAILED DESCRIPTION:
There are several forms of nonsurgical treatment for trigger finger, the most used are:

* Oral nonsteroidal and steroidal antiinflammatory's drugs use to resolve the inflammatory process
* Corticosteroids local injection: that proposes to control the inflammation, these injections have shown good effectiveness for trigger finger treatment.
* Orthotic: with the aim of to immobilize the affected joint until the resolution of the inflammatory process.
* Electrotherapeutic modalities:
* Paraffin that increases cellular metabolism and promotes peripheral vasodilatation, favoring the transduction tissue fluid, lymph flow, hyperemia and consequent absorption of exsudato.
* LASER -Lower Level Laser Therapy (LLLT): the absorption of light through the skin's photoreceptors stimulates mitochondrial chain reactions, promoting adenosine triphosphate (ATP) synthesis, acting on gene expression, which raises the level of growth factors and Tissue repair

Although the non-surgical treatment is often used there is no evidence in the literature of which is the most effective conservative treatment for trigger finger. Thus, it is necessary use appropriate methodology to define the benefits and harms of each treatment modality and assess the effectiveness of these nonsurgical treatments, and may define which one has a higher resolution and lower rates of trigger finger recurrences in short, medium and long term.

ELIGIBILITY:
Inclusion Criteria:

* 2-3 grade of trigger finger (Quinnell´s classification)
* Signing the Terms of Consent.

Exclusion Criteria:

* Presence of finger trigger in children
* Presence of traumatic finger trigger
* Secondary causes (patients with tumor of the tendon sheath,

synovitis tuberculosis, etc ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Changes in the Resolution/cure of the trigger finger until the six months of the treatment | 1, 5, 12 weeks and 6 month
  The patient must extend and flex the affected
  finger 10 times to verify the presence or absence of the trigger finger and determine
  the degree of commitment.

SECONDARY OUTCOMES:
Changes in Visual Analogue Scale (VAS) | 1, 5, 12 weeks and 6 month
Changes in Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) | 1, 5, 12 weeks and 6 month
Changes in SF-12 (quality of life) | 1, 5, 12 weeks and 6 month
Changes in the numbers of the Complications | 1, 5, 12 weeks and 6 month
Changes in the numbers of the Relapses | 1, 5, 12 weeks and 6 month

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Binder A, Hodge G, Greenwood AM, Hazleman BL, Page Thomas DP. Is therapeutic ultrasound effective in treating soft tissue lesions? Br Med J (Clin Res Ed). 1985 Feb 16;290(6467):512-4. doi: 10.1136/bmj.290.6467.512. PMID 3918652
- [Background] Colbourn J, Heath N, Manary S, Pacifico D. Effectiveness of splinting for the treatment of trigger finger. J Hand Ther. 2008 Oct-Dec;21(4):336-43. doi: 10.1197/j.jht.2008.05.001. Epub 2008 Aug 22. PMID 19006759
- [Background] Chen PT, Lin CJ, Jou IM, Chieh HF, Su FC, Kuo LC. One digit interruption: the altered force patterns during functionally cylindrical grasping tasks in patients with trigger digits. PLoS One. 2013 Dec 31;8(12):e83632. doi: 10.1371/journal.pone.0083632. eCollection 2013. PMID 24391799
- [Background] Tarbhai K, Hannah S, von Schroeder HP. Trigger finger treatment: a comparison of 2 splint designs. J Hand Surg Am. 2012 Feb;37(2):243-9, 249.e1. doi: 10.1016/j.jhsa.2011.10.038. Epub 2011 Dec 20. PMID 22189188
- [Background] Langer D, Luria S, Maeir A, Erez A. Occupation-based assessments and treatments of trigger finger: a survey of occupational therapists from Israel and the United States. Occup Ther Int. 2014 Dec;21(4):143-55. doi: 10.1002/oti.1372. Epub 2014 May 12. PMID 24821018
- [Background] Howitt S, Wong J, Zabukovec S. The conservative treatment of Trigger thumb using Graston Techniques and Active Release Techniques. J Can Chiropr Assoc. 2006 Dec;50(4):249-54. PMID 17549185
- [Background] Peters-Veluthamaningal C, van der Windt DA, Winters JC, Meyboom-de Jong B. Corticosteroid injection for trigger finger in adults. Cochrane Database Syst Rev. 2009 Jan 21;2009(1):CD005617. doi: 10.1002/14651858.CD005617.pub2. PMID 19160256
- [Background] Huisstede BM, Hoogvliet P, Coert JH, Friden J; European HANDGUIDE Group. Multidisciplinary consensus guideline for managing trigger finger: results from the European HANDGUIDE Study. Phys Ther. 2014 Oct;94(10):1421-33. doi: 10.2522/ptj.20130135. Epub 2014 May 8. PMID 24810861
- [Background] Renno AC, Toma RL, Feitosa SM, Fernandes K, Bossini PS, de Oliveira P, Parizotto N, Ribeiro DA. Comparative effects of low-intensity pulsed ultrasound and low-level laser therapy on injured skeletal muscle. Photomed Laser Surg. 2011 Jan;29(1):5-10. doi: 10.1089/pho.2009.2715. Epub 2010 Dec 18. PMID 21166589
- [Background] Salim N, Abdullah S, Sapuan J, Haflah NH. Outcome of corticosteroid injection versus physiotherapy in the treatment of mild trigger fingers. J Hand Surg Eur Vol. 2012 Jan;37(1):27-34. doi: 10.1177/1753193411415343. Epub 2011 Aug 4. PMID 21816888
- [Background] Quinnell RC. Conservative management of trigger finger. Practitioner. 1980 Feb;224(1340):187-90. No abstract available. PMID 7367373
- [Background] Valdes K. A retrospective review to determine the long-term efficacy of orthotic devices for trigger finger. J Hand Ther. 2012 Jan-Mar;25(1):89-95; quiz 96. doi: 10.1016/j.jht.2011.09.005. PMID 22265444
- [Background] Dingemanse R, Randsdorp M, Koes BW, Huisstede BM. Evidence for the effectiveness of electrophysical modalities for treatment of medial and lateral epicondylitis: a systematic review. Br J Sports Med. 2014 Jun;48(12):957-65. doi: 10.1136/bjsports-2012-091513. Epub 2013 Jan 18. PMID 23335238
- [Background] Dilek B, Gozum M, Sahin E, Baydar M, Ergor G, El O, Bircan C, Gulbahar S. Efficacy of paraffin bath therapy in hand osteoarthritis: a single-blinded randomized controlled trial. Arch Phys Med Rehabil. 2013 Apr;94(4):642-9. doi: 10.1016/j.apmr.2012.11.024. Epub 2012 Nov 24. PMID 23187044
- [Background] Sibtain F, Khan A, Shakil-Ur-Rehman S. Efficacy of Paraffin Wax Bath with and without Joint Mobilization Techniques in Rehabilitation of post-Traumatic stiff hand. Pak J Med Sci. 2013 Apr;29(2):647-50. PMID 24353596
- [Background] Beaton DE, Wright JG, Katz JN; Upper Extremity Collaborative Group. Development of the QuickDASH: comparison of three item-reduction approaches. J Bone Joint Surg Am. 2005 May;87(5):1038-46. doi: 10.2106/JBJS.D.02060. PMID 15866967
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- See also: World Association of Laser Therapy. Recommended antiinflammatory dosage for low level laser therapy. 2005. (accessed june 20, 2017). — http://www.walt.nu/dosage-recommendations.html